CLINICAL TRIAL: NCT00674076
Title: Clinical Application of Ultrasound in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200802028R
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- sleep apnea: a patient has been diagnosed as having obstructive sleep apnea
- control: a case who has a negative polysomography or noraml score of Pittsburg sleep questionaire

SUMMARY:
We hypothesize the width air-colum of retropalatal region and tongue voulme by ultrsound through submental area is different between normal control with those with obstructive sleep apnea syndrome who was comfirmed by polysomography.

DETAILED DESCRIPTION:
Patients with obstructive sleep apnea mainly due to upper airway narrowing are evaluated conventionaly by polysomography. Recently, the magnetic resonace imaging has been well established in evaluating upper airway and correlating with the severity by tongue mass and the area of retropalatal airway. However, some drawbacks of MRI includes expensiveness might lead its less use. As for ultrasound which is very popularly applied in medical illness, is more convenient and money saving than MRI. We propose that ultrsound measuring the tongue volume and width of upper airway through submental area may be a alternative image for a upper airway measuring.

ELIGIBILITY:
Inclusion Criteria:

* group of sleep apnea: patients who have been diagnosed as having obstructive sleep apnea
* control group: patients who have a negative polysomogrphy or a normal score of Pittsburg sleep questionaire

Exclusion Criteria:

* Less than 18-year-old
* un-willing
* not co-operated person

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who are arranged to recived polysomography
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | less than one month apart from ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chien Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital, Internal Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Shu CC, Lee P, Lin JW, Huang CT, Chang YC, Yu CJ, Wang HC. The use of sub-mental ultrasonography for identifying patients with severe obstructive sleep apnea. PLoS One. 2013 May 10;8(5):e62848. doi: 10.1371/journal.pone.0062848. Print 2013. PMID 23675433